CLINICAL TRIAL: NCT02710162
Title: Determination of Accurate Screening Tools for Dysphagia in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Accurate Screening Tools for Dysphagia in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201600163
Record Dates: First submitted 2016-02-29; First posted 2016-03-16 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Capsaicin; Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening (Experimental): Participants enrolled will have the following test: Micro Mouth Pressure Meter, reflexive cough testing (with capsaicin used in blocks), lingual strength and endurance trials using the Iowa Oral Performance Instrument, Electrical Impedance Myography of the tongue, Pulmonary Function Testing, and a Videofluoroscopic Swallowing Study. In addition, the patient will complete the following surveys: Swallowing Related Quality of Life Questionnaire (SWAL-QOL), Eating Assessment Tool-10 (EAT-10), Functional Oral Intake Scale (FOIS), Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R), The Center for Neurologic Studies Bulbar Function Scale (CNS-BFS), and the Communicative Effectiveness Survey (CES).
  Interventions: Device: Micro Mouth Pressure Meter; Device: Iowa Oral Performance Instrument; Device: Electrical Impedance Myography; Drug: Capsaicin; Procedure: Videofluoroscopic Swallowing Study; Procedure: Pulmonary Function Testing; Other: Swallowing Related Quality of Life Questionnaire; Other: Functional Oral Intake Scale; Other: Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised; Other: Eating Assessment Tool-10; Other: Communicative Effectiveness Survey; Other: The Center for Neurologic Studies Bulbar Function Scale

INTERVENTIONS:
Device: Micro Mouth Pressure Meter — The participant will be seated with the nose occluded using a nose clip. After inhaling to total lung capacity, the participant will place his or her lips around the mouthpiece and blow out as forcefully as possible. A flanged rubber mouthpiece will be used to overcome the inability of some individuals to create tight lip seal due to facial muscle weakness. Three trials will be performed and the patients highest maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) used.
  Other Names: digital manometer; Micro medical device
Device: Iowa Oral Performance Instrument — The Iowa Oral Performance Instrument (IOPI) is a device that measures the peak pressure performance of lingual strength and endurance via the action of a bulb placed on the hard palate.
  Other Names: IOPI
Device: Electrical Impedance Myography — The SFB7 Bioimpedance device measures the function of the tongue by calculating measures of reactance, resistance and phase once a custom electrode array is placed on the midline of the subject's tongue for approximately 2 seconds.
  Other Names: EIM
Drug: Capsaicin — A capsaicin challenge with three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin. The capsaicin will be dissolved in a vehicle solution consisting of 80% physiological saline, and 20% ethanol. Participants will be given the instruction "cough if you need to" prior to capsaicin delivery.The solution will be administered automatically upon detection of an inspired breath and there will be a minimum of one minute between each trial. This is to test the reflexive cough testing for upper airway sensitivity and motor thresholds.
  Other Names: Hot pepper
Procedure: Videofluoroscopic Swallowing Study — Videofluoroscopic swallowing study will be performed to measure the oropharyngeal swallowing.
  Other Names: VFSS; modified barium swallow (MBS); X-Ray of swallowing
Procedure: Pulmonary Function Testing — Pulmonary Function testing will be performed using conventional methods and will include the following outcomes: forced vital capacity (FVC), sniff nasal inspiratory pressure (SNIP), peak expiratory flow (PEF), forced expiratory volume (FEV1) expressed as a percentage of predicted values.
Other: Swallowing Related Quality of Life Questionnaire — Swallowing Quality of Life Questionnaire (SWAL-QOL) will be used for participant reporting of swallow-related quality of life.
  Other Names: SWAL-QOL
Other: Functional Oral Intake Scale — The Functional Oral Intake Scale (FOIS) will be used for participants to report their food intake habits.
  Other Names: FOIS
Other: Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised — The Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) will be used to track global disease progression in participants.
  Other Names: ALSFRS-R
Other: Eating Assessment Tool-10 — The Eating Assessment Tool-10 will be used for participant reporting of swallowing system severity.
  Other Names: EAT-10
Other: Communicative Effectiveness Survey — The Communication Effectiveness Survey (CES) will be used for participant reporting of communication abilities across different speech contexts.
  Other Names: CES
Other: The Center for Neurologic Studies Bulbar Function Scale — The Center for Neurologic Studies Bulbar Function Scale (CNS-BFS) will be used to report bulbar function in study participants.
  Other Names: CNS-BFS

SUMMARY:
Individuals with th Amyotrophic Lateral Sclerosis are at high risk for swallowing impairment (dysphagia) which leads to malnutrition, decreased pulmonary health, aspiration and aspiration pneumonia. These sequelae necessitate timely identification of at risk individuals to ensure optimal management of oral intake and pulmonary function. The purpose of this study is to evaluate the discriminant ability of several non-invasive screening tools at detecting swallowing impairment in individuals with ALS.

DETAILED DESCRIPTION:
This research study is being performed to determine how accurate different screening tools or tests are at identifying swallowing problems associated with Amyotrophic Lateral Sclerosis (ALS).

As a participant one evaluation will be performed at the University of Florida Swallowing Systems Core laboratory located at Shands Hospital, Gainesville will take place. This will take approximately two-hours. During this evaluation an videofluoroscopy (X-ray of swallowing), cough tests, tongue function test and questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable or definite ALS

Exclusion Criteria:

* allergies to barium or capsaicin
* tracheotomy or mechanical ventilation
* absence of diaphragmatic pacer
* respiratory disease (COPD).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
The Penetration-aspiration scale will be used to measure swallowing function | Baseline
The IOPI will be used to measure Lingual strength and endurance | Baseline
  The Iowa Oral Pressure Instrument device will measure the peak performance of lingual strength a via the action of a bulb placed on the hard palate. To assess maximum anterior isometric pressure, the bulb will be placed on the roof of the mouth and the participant will raise his or her tongue to apply pressure to this bulb and then quickly release the tongue back into a neutral position. This repetitive tongue movement will be performed three times and values will be recorded.
The oral pneumatograph will be used to measure voluntary cough function | Baseline
  Voluntary cough function will be assessed using an oral pneumotachograph, connected to a spirometer filter during voluntary cough production. The participant will be seated with a respiratory face-mask held in place by the examiner and instructed to complete three tidal breaths into the face-mask, airflow signal will be measured
The nebulizer with cough protocol will be used to measure reflexive cough | Baseline
  Reflexive cough will be assessed using an oral pneumotachograph, differential pressure transducer, and have a side port with a one-way inspiratory valve for nebulizer connection. The nebulizer will deliver three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin.

SECONDARY OUTCOMES:
Global disease progression as confirmed by the ALS Functional Rating Scale-Revised (ALSFRS-R) | Baseline
  The ALSFRS-R includes 12 questions. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 48=best.
Participant perception of swallowing impairment as confirmed by Swallowing Quality of Life Questionnaire (SWAL-QOL) | Baseline
  SWAL-QOL is a standardized psychometric scale measuring swallow-related QOL and containing 44-items relating to swallowing specific quality of life measured across 10 domains. Individual domain scores and a total SWAL-QOL score will be derived. Scores range from 0 to 100, with a score of 100 representing no impairment (the most favorable state)
Dietary intake as confirmed by Functional Oral Intake Scale (FOIS) | Baseline
  FOIS is a validated 7-point scale indexing an individual's ability to intake food on a day-to-day basis.
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Participant perception of swallowing related symptoms as confirmed by The Eating Assessment Tool 10 (EAT-10) | Baseline
  EAT-10 is a 10-item validated self-administered dysphagia severity symptom survey. Score is 0 - 40 with 0 being the best possible score and 40 the worst possible score.
Participant perception of communication abilities as confirmed by Communication Effectiveness Survey | Baseline
  A measure of self-rated communication abilities across a variety of settings as perceived by the patients and/or their caregivers will be measured using the 8-point Communication Effectiveness Survey (CES)
Bulbar function confirmed by the Center for Neurologic Studies Bulbar Function Scale (CNS-BFS) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No